## In the Patient's Words: Understanding Patient Participation and Engagement in Plaque Psoriasis Clinical Trials

Presented is the informed consent form for participants diagnosed with plaque psoriasis who are enrolling in <a href="Power Clinical Trial's">Power Clinical Trial's</a> observational clinical study.

Date: March 22, 2024

Introduction to the Study

You're invited to participate in our research initiative. This document acts as a consent form, offering insights into the study and its potential impact on you. If you come across any unclear terms or phrases, feel free to seek clarification from our research team. We encourage you to take your time considering your participation and ask any questions you may have. It may be helpful to discuss the study with your loved ones, personal physician, trusted healthcare providers, or community members. Remember, participation in this study is voluntary, and you're under no obligation to join.

Understanding Plaque Psoriasis: Overview of an Observational Study

The objective of this study is to observe and comprehend various factors influencing the process of enrolling in and completing your plaque psoriasis clinical trial.

Collected data will be anonymized and analyzed to identify trends in the experiences of plaque psoriasis patients, which often impact enrollment rates or trial completion.

Since this clinical study is observational, there will be no changes to your treatment upon participation.

This document serves as written confirmation of discussions with our site staff or recruitment coordinators and can be used as a reference during your participation in this clinical study.

Investigating the Purpose of Plaque Psoriasis Research

Clinical trials tend to favor particular demographic groups, yet there is a lack of research explaining which trial attributes impact participation.

This study aims to collect a broad spectrum of data on the clinical trial experiences of plaque psoriasis patients to determine which factors hinder a patient's ability to enroll in or complete a trial.

Additionally, it seeks to analyze data from different demographic perspectives to identify recurring trends that may offer insights for the benefit of future plaque psoriasis patients.

Understanding the Advantages of Joining This Clinical Study

Your participation in this observational clinical trial is essential for uncovering ways to support future plaque psoriasis patients more effectively. The insights gained may lead to improvements in participation rates and expand the impact of future studies.

Understanding the Risks of Participating in This Observational Clinical Study

Engaging in clinical trials may necessitate alterations to your treatment routines, which inherently carry certain risks.

However, as this is an observational clinical study, there will be no modifications to your treatment regimen, thus eliminating any associated risks related to treatment changes.

Throughout the trial, online reporting and video calls with participating plaque psoriasis patients are utilized. One potential risk in this process is the potential for data breaches.

With Power's clinical trials, this risk is mitigated. We ensure that data shared during these calls is securely encrypted. Call logs and electronic copies of consent forms are stored anonymously in a highly secure environment.

Exploring Potential Risks in This Observational Clinical Study

Participation in clinical trials may involve adjustments to your treatment protocols, which inherently carry certain risks.

However, since this is an observational clinical study, there will be no modifications to your treatment regimen, thus eliminating any associated risks stemming from treatment changes.

Throughout the trial, online reporting and video calls with participating plaque psoriasis patients are utilized. One potential risk in this process is the potential for data breaches.

With Power's clinical trials, we prioritize security to minimize this risk. We ensure that data exchanged during these calls is securely encrypted. Call logs and electronic copies of consent forms are stored anonymously in a highly secure environment.

Unique Aspects of This Research Compared to Other Plaque Psoriasis Clinical Trials

In contrast to many other trials, this study does not involve intervention.

Interventional clinical trials typically require plaque psoriasis patients to undergo a prescribed treatment regimen, potentially different from their current one.

However, as an observational clinical trial, there will be no alterations to your treatment in this study.

If you're interested in exploring other studies, you can search for <u>plaque psoriasis</u> <u>studies</u> on clinicaltrials.gov or <u>plaque psoriasis clinical trials</u> on Power's website.

Delve deeper into clinical trials and their enrollment rates by exploring the following sources:

Oyer, Randall A., Patricia Hurley, Leigh Boehmer, Suanna Steeby Bruinooge, Kathryn Levit, Nadine Barrett, Al Benson et al. "Increasing racial and ethnic diversity in cancer clinical trials: an American Society of Clinical Oncology and Association of Community Cancer Centers joint research statement." *Journal of Clinical Oncology* 40, no. 19 (2022): 2163-2171.

Cooper, Richard S., and Bruce M. Psaty. "Diversity and inclusiveness should remain the guiding principles for clinical trials." *Circulation* 112, no. 23 (2005): 3660-3665.

## Requirements for Plaque Psoriasis Patients in This Study

In this study, participants are expected to complete bi-weekly surveys, each lasting around 30 minutes. Additionally, quarterly check-in calls will be scheduled throughout the clinical trial period.

To enroll, individuals must currently be participating in an interventional clinical trial. Joining this observational study will not alter the treatment or methodology prescribed by their primary care physician.

Throughout the trial duration, participants should promptly address any concerns or questions by contacting our staff for clarification.

Prior to enrolling in this clinical study, individuals are required to consult with their care team.

## Participant Acknowledgment

I have carefully read and understood the information presented above, and it has been verbally explained to me in detail. All my queries have been satisfactorily answered.

I recognize that my involvement in this observational study is entirely voluntary, and I reserve the right to withdraw at any time. Signing this form does not waive any of my legal rights.

I understand that I will be provided with a copy of this consent form. By signing below, I am indicating my intention to participate in the clinical study.

| Printed Name of Participant | |
|---|---|
| Participant Signature | |
| Date | |
| Verification of Informed Consent Dis | cussion |
| I affirm that I have meticulously gone throuparticipant. | ugh the contents of this form with the |
| I guarantee that the participant has a clear understanding of the benefits, risks, and procedures related to this clinical trial focusing on plaque psoriasis. | |
| Printed name of Person Conducting Inforn | ned Consent Discussion |
| Person Conducting Informed Consent Discussion Signature | |
| Date | |